CLINICAL TRIAL: NCT03882437
Title: A Clinical Study Evaluating a Recombinant Adeno-Associated Virus Serotype 9 (rAAV9) Capsid Containing the Human Lysosome-Associated Membrane Protein 2 Isoform B (LAMP2B) Transgene (RP-A501; AAV9.LAMP2B) in Male Patients With DD
Brief Title: Gene Therapy for Male Patients With Danon Disease (DD) Using RP-A501; AAV9.LAMP2B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-A501-0219
Record Dates: First submitted 2019-03-12; First posted 2019-03-20 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Danon Disease
Keywords: hypertrophic cardiomyopathy; HCM; X-linked disease; LAMP 2A; Pediatric; Skeletal myopathies
MeSH Terms: conditions — Glycogen Storage Disease Type IIb; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Evaluation of RP-A501 in pediatric patients (ages 8-14) will commence only pending determination of safety in the older (adult and age 15-17) population.
  In Phase 1, RP-A501 will be investigated in three treatment cohorts, as follows with a single cohort currently recruiting:
  Cohort 1: Adult and age 15-17: 6.7 × 1013 GC/kg (n=3-4)
  Cohort 2: Adult and age 15-17: 1.1 × 1014 GC/kg (n=2 [patients already treated; closed for current enrollment])
  Cohort 1A: Pediatric age 8-14: 6.7 × 1013 GC/kg (n=2-4)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-A501 (Experimental): RP-A501 is a gene therapy product consisting of a rAAV9 capsid containing the human LAMP2B transgene which will be administered as a single intravenous (IV) infusion. Subjects will receive one of three dose levels depending on the cohort.
  Interventions: Biological: RP-A501

INTERVENTIONS:
Biological: RP-A501 — RP-A501 is a gene therapy product consisting of a rAAV9 capsid containing the human LAMP2B transgene which will be administered as a single IV infusion.

SUMMARY:
This is a non-randomized open-label Phase 1 study to evaluate the safety and toxicity of gene therapy using a recombinant adeno-associated virus serotype 9 (AAV9) containing the human lysosome-associated membrane protein 2 isoform B (LAMP2B) transgene (investigational product (IP), RP-A501) in male patients with Danon Disease (DD).

DETAILED DESCRIPTION:
The study is a non-randomized open-label Phase I clinical trial to characterize the safety and toxicity associated with infusion of a recombinant adeno-associated serotype 9 (rAAV9) capsid containing the human lysosome-associated membrane protein 2 isoform B (LAMP2B) transgene (investigational product (IP), RP-A501) in male patients with Danon Disease (DD).

During the course of the study, approximately 7-10 male subjects age 8 and over will receive a single intravenous (IV) infusion of the IP. Prior to infusion of IP, rituximab and sirolimus will be administered prophylactically.

All patients are planned to be followed for 36 months after investigational product administration. After the end of the follow-up period, patients will enter a Long-Term Follow-Up (LTFU) study enabling follow-up for an additional 2 to 5 years post-IP administration.

The study will also enable an initial evaluation of whether or not the IP results in cardiomyocyte and skeletal muscle transduction and gene expression and preliminary assessment of the extent of cardiomyocyte and histologic correction. Additionally, a preliminary evaluation of clinical stabilization following infusion will also be made.

ELIGIBILITY:
Main Criteria for Inclusion:

The study will enroll adult and pediatric males with a confirmed diagnosis of DD. Patients may be of any race or ethnicity. Patients and/or competent custodial parents must provide informed written consent and meet all of the enrollment criteria as detailed subsequently to be eligible to participate.

1. DD diagnosis with any confirmed LAMP2 mutation(s).
2. Cardiac involvement as documented by at least one abnormal finding on electrocardiogram (ECG), echocardiogram, gadolinium-enhanced cardiac magnetic resonance imaging (MRI), or electrophysiology study.
3. Age ≥15 years for cohorts 1 and 2; 8-14 years for cohorts 1A.
4. Male gender.
5. New York Heart Association (NYHA) Class II or III.
6. Adequate hematologic function as defined by hemoglobin, absolute neutrophil count (ANC), and platelet count ≥ lower limit of normal (LLN).
7. Adequate hepatic function as defined by:

   1. AST and ALT ≤10.0×ULN or GGT ≤2.0×ULN (transaminase elevations in DD are considered extensively to result from muscle injury; hence the relatively high upper limit for transaminases and consideration of GGT level, and the presence of additional hepatic eligibility markers of bilirubin and PT/INR).
   2. Serum bilirubin ≤1.2×ULN (i.e., Grade ≤1 bilirubin increase).
   3. PT/INR ≤1.2×ULN (in the absence of anticoagulation).
   4. Absence of cirrhosis or other signs of inflammation on liver ultrasound
8. Adequate renal function as defined by creatinine ≤ULN.
9. Ability to provide informed consent (for adult patients and parents/legal guardians of pediatric patients) and assent (for patients age 15-17).
10. Ability to comply with study procedures including investigational therapy and follow-up evaluations.
11. Able to walk >150 meters unassisted during the 6MWT.
12. Patient has received meningococcal vaccination recommended by Centers for Disease Control as appropriate for age and health condition (vaccination must be performed at least 6 weeks prior to IP administration).

Main Criteria of Exclusion:

Patients meeting any of the following criteria are not eligible for study participation:

1. I.V. therapy with positive inotropes, vasodilators, or diuretics within the 30 days prior to enrollment (i.e., patient must be stable on oral medical therapy).
2. Prior cardiac transplantation or prior transplant of other organ (lung, liver, other).
3. Prior cardiac surgery and/or percutaneous cardiac intervention for arteriothrombotic complications, or valvuloplasty.
4. Presence or requirement of a Left Ventricular Assisted Device (LVAD).
5. History of intracardiac thrombosis or arteriothromboembolic events including stroke or transient ischemic attack (TIA).
6. Left ventricular ejection fraction (LVEF) <40% at baseline.
7. History of the following prior arteriothromboembolic complications: myocardial infarction or unstable angina.
8. Significant (greater than moderate) valvular stenosis or regurgitation on echocardiogram.
9. Requires mechanical ventilation.
10. Anti-AAV9 neutralizing antibody titer >1:40.
11. Concurrent enrollment in any other clinical investigation involving use of an investigational agent for the treatment of CHF or cardiomyopathy.
12. Active hepatitis B or C infection (including patients with positive hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis B core antibody (HBcAb), or detectable hepatitis B virus (HBV) or hepatitis C virus (HCV) viral load). Patients with previous, adequately resolved HBV or HCV are eligible.
13. Significant medical conditions including documented human immunodeficiency virus (HIV) infection, active viral or other hepatitis, poorly-controlled hypertension or diabetes, poorly controlled cardiac arrhythmia, or uncontrolled viral, bacterial, or fungal infection.
14. Any concomitant medical or psychiatric condition that in the opinion of the Investigator renders the patient unfit for study participation or at higher than acceptable risk for study participation.
15. Active hematologic or solid organ malignancy, not including non-melanoma skin cancer or other carcinoma in situ. Patients with previously resected solid organ malignancies or definitively treated hematologic malignancies may be eligible if there has been no evidence of active malignancy during the prior 3 years.
16. Any contraindication to use of sirolimus which includes hypersensitivity to sirolimus or HC-60 (polyoxyl 60 hydrogenated castor oil).
17. Active or latent tuberculosis.

Min Age: 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by United States (US) National Cancer Institute Common Terminology Criteria (NCI CTCAE) | 3 years
  Evaluation of safety associated with RP-A501
Number of participants within each dose level cohort with treatment-related adverse events as assessed by United States (US) National Cancer Institute Common Terminology Criteria (NCI CTCAE) | 3 years
  Assessment of safety at both doses (single IV administration)
Evaluation of cardiomyocyte histologic correction following administration of RP-A501 via endomyocardial biopsy | 3 years
  Assessment of cardiomyocyte histologic correction following administration of RP-A501 via endomyocardial biopsy
Preliminary evaluation of clinical stabilization of cardiomyopathy following administration of RP-A501 via cardiopulmonary testing | 3 years
  Assessment of clinical stabilization of cardiomyopathy following infusion of RP-A501 via cardiopulmonary testing

SECONDARY OUTCOMES:
Determination of the percentage of patients in whom RP-A501 resulted in a sustained improvement or stabilization in cardiovascular pathophysiology | 3 years
  Evaluation of sustained improvement or stabilization in cardiovascular pathophysiology as assessed by medical evaluation, radiographic evaluation of cardiac structure and function, and cardiopulmonary exercise/physiologic parameters
Determination of the percentage of patients in whom cardiomyocytes corrected LAMP2B gene and/or protein | 3 years
  Evaluation of the percentage of patients in whom cardiomyocytes contain the corrected LAMP2B gene and/or protein and improvement in DD-associated histologic abnormalities and when feasible to quantify the extent of genetic and histologic correction in the myocardium.
Determination and characterization of immunologic response to RP-A501 | 3 years
  Assessment of potential immunogenicity to the components of the investigational product
Determination of the percentage of patients who require and/or receive treatment for heart failure following RP-A501 | 3 years
  Assessment of the percentage of patients who require and/or receive subsequent cardiac transplantation, left ventricular assist device (LVAD), implantable cardioverter-defibrillator or pacemaker placement, electrophysiologic ablative procedure for cardiac conduction aberrancy or subsequent hospitalizations for heart failure.
Evaluation of overall survival | 3 years
  Assessment of overall survival post RP-A501

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rossano, MD, Principal Investigator — Children's Hospital of Philadelphia; Matthew Taylor, MD, PhD, Principal Investigator — University of Colorado, Anschutz Medical Ctr; Barry Greenberg, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - University of Colorado, Aurora, Colorado
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Greenberg B, Taylor M, Adler E, Colan S, Ricks D, Yarabe P, Battiprolu P, Shah G, Patel K, Coggins M, Carou-Keenan S, Schwartz JD, Rossano JW. Phase 1 Study of AAV9.LAMP2B Gene Therapy in Danon Disease. N Engl J Med. 2025 Mar 6;392(10):972-983. doi: 10.1056/NEJMoa2412392. Epub 2024 Nov 18. PMID 39556016
- [Derived] Grisorio L, Bongianino R, Gianeselli M, Priori SG. Gene therapy for cardiac diseases: methods, challenges, and future directions. Cardiovasc Res. 2024 Nov 25;120(14):1664-1682. doi: 10.1093/cvr/cvae207. PMID 39302117
- [Derived] O'Neil EC, Uyhazi KE, O'Connor K, Aleman IA, Pulido JS, Rossano JW, Aleman TS. DANON DISEASE: A MODEL OF PHOTORECEPTOR DEGENERATION SECONDARY TO PRIMARY RETINAL PIGMENT EPITHELIUM DISEASE. Retin Cases Brief Rep. 2022 Nov 1;16(6):707-713. doi: 10.1097/ICB.0000000000001125. PMID 36288619